CLINICAL TRIAL: NCT02774447
Title: Day-Case Closure of Ileostomy: A Pilot Study
Brief Title: Day-Case Closure of Loop Ileostomy in Rectal Cancer
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: Dnr 2014/363
Record Dates: First submitted 2015-09-28; First posted 2016-05-17 (Estimated); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Ileostomy Closure in Rectal Cancer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rectal cancer patients with ileostoma: In association with anterior resection of rectal cancer these patients obtain loop-ileostoma in order to avoid complications. These are closed within a few months and according to previous studies the admission time is 3-5 days after operation. This study is a single-arm study. The arm include patients having had rectal cancer operation and who have obtained a loop-ileostoma and that meet the inclusion criteria.
  The operation procedure is standardized; shortly described by dissecting the ileostoma from the abdominal wall and everting the stoma ledges, which will be sutured or stapled. The patients will be observed for 23 hours, and if there are no contraindications according to described criteria the patient can be discharged form the hospital, however all patients will be followed up.
  Interventions: Procedure: ileostoma closure

INTERVENTIONS:
Procedure: ileostoma closure — The operation procedure is standardized as described above (see group description).The patients will be observed for 23 hours, and if there are no contraindications according to described criteria the patient can be discharged form the hospital, however all patients will have follow-up telephone contact on a daily basis with a nurse for the first week. Patients will meet the surgeon 3 days after discharge and after 4 weeks.

SUMMARY:
The aim of this study is to investigate if day-case closure of ileostomy is feasible and safe.

DETAILED DESCRIPTION:
For all patients that match the inclusion criteria a registration-protocol is completed. Then the patients are operated and a surgery-protocol is completed. The patients are observed for maximum 24 h and discharged if they meet the discharge-criteria. 30 days post-operative the investigators do a follow-up of complications.

ELIGIBILITY:
Inclusion Criteria:

* Adults not older than 80 planed for closure of ileostomy
* The patient should not have had the ileostomy for more than 1 year
* Informed written consent should be given
* The patient should have a phone
* Should have an adult supervision at home for the first 24 hours after discharge
* American Society of Anesthesiologists (ASA) classification 1-2

Exclusion Criteria:

* ASA classification 3 and above
* The pre-operative investigation have shown anastomosis leakage or stricture
* Dementia or other cognitive dysfunction
* The need of an interpreter
* Patients assessed not being able to manage themselves at home post-operative
* Insulin treated diabetes
* Coagulopathy
* Other organ dysfunction
* Bleeding more than 300 ml
* If converted to laparatomy
* Other intraoperative difficulties leading to suspected increased risk of complication

Discharge criteria:

* Stable vital parameters regarding circulation and respiration
* No sign of bleeding
* Pain relief possible through per oral administration
* Emptied urinary bladder
* Able to maintain per oral nutrition
* Mobilization possible
* Obtained oral and written information about symptoms of sepsis and bowel obstruction
* Obtained telephone number of a contact-nurse
* Obtained time for wound-inspection at the surgical unit

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients earlier operated at the local hospital, who are now planned for closure of ileostomy
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-08; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Number of patients with complications | 30 days
Number of patients re-admitted | 30 days
Number of patients re-operated | 30 days
Number of patients who were able to return home after day-case closure of loop-ileostomy | 24 houres

CONTACTS AND LOCATIONS:
Overall Officials: Abbas Chabok, Phd, MD, Study Director — Centrum for Clinical Research Västerås/Uppsala University
Locations (1):
- Landstinget Västmanland,Centrum för klinisk forskning, Västerås, Sweden

REFERENCES:
- [Derived] Afshari K, Nikberg M, Smedh K, Chabok A. Loop-ileostomy reversal in a 23-h stay setting is safe with high patient satisfaction. Scand J Gastroenterol. 2021 Sep;56(9):1126-1130. doi: 10.1080/00365521.2021.1947367. Epub 2021 Jul 5. PMID 34224302